CLINICAL TRIAL: NCT06683755
Title: Phase I/IIa Dose Finding Study of Triplet Regimen of Relatlimab Ipilimumab and NIvolumab in First Line Therapy of Metastatic Melanoma (TRINITY)
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1032; NCI-2024-09421 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; relatlimab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Phase I + IIa: Nivolumab + Relatlimab + Ipilimumab (Experimental): Participants particiapting on study will be randomized
  Interventions: Drug: Nivolumab; Drug: Relatlimab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — Given by IV
Drug: Relatlimab — Given by IV
Drug: Ipilimumab — Given by IV

SUMMARY:
To determine the recommended Phase IIa dose (RP2D) of the triplet combination.

To determine the safety and efficacy of the combination at the RP2D.

DETAILED DESCRIPTION:
Primary Objectives:

Phase I:

Primary Objective of the Phase I portion is to determine the recommended Phase IIa dose (RP2D) of ipilimumab in combination with nivolumab and relatlimab in the first line treatment of patients with metastatic melanoma.

Phase IIa:

Primary Objective of the Phase IIa portion is to determine the preliminary clinical efficacy of ipilimumab at the RP2D in combination with nivolumab and relatlimab in the first line treatment of patients with metastatic melanoma as determined by overall response rate (ORR) according to RECIST 1.1.

Secondary Objectives:

1. Phase I: To assess the overall response rates by RECIST 1.1 (as assessed by Investigator/site designated radiologist).
2. Phase IIa: To determine the safety and tolerability of the triplet combination.
3. To assess the progression free survival (PFS), and overall survival for patients treated with the triplet combination
4. Assess the PFS and ORR to subsequent therapies in the second and third line setting.
5. Evaluate the pharmacodynamic effects of the combination in tumor tissues obtained at baseline (archival and/or fresh tissue), on treatment, and at time of progression.
6. Peripheral blood assays to assess for immunologic changes and immune cell subsets

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. ECOG performance status 0-1
3. Subjects must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol-related procedures that are not part of normal subject care.

   • Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study.
4. Histologically confirmed unresectable stage III or stage IV malignant melanoma (Stage IV).
5. At least one measurable target lesion according to RECIST 1.1. (Appendix 1), which previously was not treated.

   • Growth or change in a lesion previously irradiated will not be considered measurable. Regrowth in cavity of previously excised lesion will not be considered measurable
6. Tumor tissue from an unresectable or metastatic site of disease must be available for biomarker analyses. The biopsy should be a core biopsy, a punch biopsy, an excisional biopsy, or a surgical specimen. Fine needle aspiration is unacceptable for submission

   * For Phase I participants: Pretreatment tissue must be available through either an archival sample obtained within at most 6 months and submitted as an FFPE tissue block or 30 unstained tumor tissue slides or a fresh pretreatment biopsy. Subsequent tumor biopsies will be optional.
   * For Phase IIa participants: Either an archival sample submitted as an FFPE tissue block or unstained tumor tissue slides or a fresh pretreatment biopsy from safely biopsiable lesion. Note that if the patient has archival tissue available from a biopsy within 90 days of C1D1 and there has been no systemic treatment since that time then that tissue can be used in place of a fresh pre-treatment biopsy. Patients must also agree to undergo post treatment, cycle 2, tumor biopsies for research purposes. Subsequent biopsies will be optional.
7. No prior systemic lines of treatment for metastatic melanoma. Prior adjuvant or neo-adjuvant therapy will be permitted as long as it did not contain ipilimumab and the last dose has been >6 months.
8. Prior radiation is allowed with a two week wash out period prior to initiation of treatment.
9. Adequate organ function as described below.

   Table 2. Evaluation of Organ Function Laboratory Value Hematological Absolute neutrophil count (ANC) ≥ 1.5 X 109/L Platelets ≥ 100 X 109/L (≥ 60 for HCC) Hemoglobin ≥ 8.0 g/dL Renal Creatinine OR ≤1.5 × ULN OR Measured or calculatedb creatinine clearance ≥40 mL/min for participant with creatinine levels >1.5 × institutional (GFR can also be used in place of creatinine or ULN CRCl) Hepatic ≤1.5 ×ULN OR direct bilirubin ≤ULN Total bilirubin for participants with total bilirubin levels AST (SGOT) and ALT (SGPT) ≤3.0 × ULN (≤5 × ULN for participants with liver metastases) Coagulation International normalized ratio (INR) OR ≤1.5 × ULN unless participant is receiving prothrombin time (PTT) anticoagulant therapy as long as PT or Activated partial thromboplastin time aPTT wi withing therapeutic range of intended use of anticoagulants (aPTT) ALT (SGPT)=alanine aminotransferase (serum glutamic pyruvic transaminase); AST (SGOT)=aspartate aminotransferase (serum glutamic oxaloacetic transaminase); GFR=glomerular filtration rate; ULN=upper limit of normal.

   a Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks.

   b Creatinine clearance (CrCl) should be calculated per institutional standard. NOTE: This table includes eligibility-defining laboratory value requirements for treatment; laboratory value requirements should be adapted according to local regulations and guidelines for the administration of specific chemotherapies.
10. Women of child-bearing potential (WOCBP) must not be breastfeeding and must have a negative pregnancy test within 3 days prior to initiation of dosing. She must agree to use an acceptable method of birth control from the time of the negative pregnancy test, through the duration of treatment with the study combination plus 5 half-lives of study treatment for a total of 5 months post -treatment completion. WOCBP must agree to adhere to the contraceptive guidance in Appendix 4. NOTE: A female participant is eligible to participate if she is not a woman of childbearing potential as defined Appendix 4.
11. All associated toxicity from previous or concurrent cancer therapy must be resolved (to ≤ grade 1 or baseline) prior to study treatment administration. This excludes low grade or non-serious toxicities. However, stable endocrinopathies requiring replacement therapy will be allowed.
12. Steroids for physiological replacement are allowed as long as it does not exceed 10 mg/day prednisone equivalents.
13. Participants must have known BRAF V600 mutation status or consent to BRAF V600 mutation testing per local institutional standards during the screening period. BRAF V600 results need not be available at the time of study start.
14. Participants with asymptomatic brain metastases are eligible. There must also be no requirement for immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalents) for at least 10 days prior to study treatment administration. Patients with brain metastases treated with SRS will be allowed, as long as last radiation therapy is >1 week.

Exclusion Criteria:

1. Patients with ocular melanoma.
2. Patients with symptomatic CNS metastases and/or requiring corticosteroid treatment.
3. History of known leptomeningeal involvement (lumbar puncture not required).
4. Patients who experienced Grade 3/4 immune-related adverse events with checkpoint inhibitor therapy, except those that are unlikely to re-occur with standard countermeasures (e.g. hypothyroidism) 5. Subjects with an active, known or suspected autoimmune disease. Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.

6. Subjects with major medical, neurologic or psychiatric condition who are judged as unable to fully comply with study therapy or assessments should not be enrolled.

7. Subject has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years. Note: The time requirement does not apply to participants who underwent successful treatment of superficial bladder cancer, in situ cervical cancer, or other in-situ cancers. Subjects with a completely treated prior malignancy and no evidence of disease for ≥ 2 years are eligible.

a. Skin Cancer Exclusion: Please note that basal cell carcinoma and squamous cell carcinoma is exempt from needing resection prior to treatment. (Resection can be completed after the start of treatment).

8. History of or is positive for hepatitis B (hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (hepatitis C virus [HCV] RNA [qualitative] is detected).

a. NOTE: Without known history, testing needs to be performed to determine eligibility. Hepatitis C antibody (Ab) testing is allowed for screening purposes in countries where HCV RNA is not part of standard of care.

9. History of human immunodeficiency virus (HIV) infection. No HIV testing is required unless mandated by local health authority.

10. The use of corticosteroids is not allowed for 14 days prior to initiation of therapy (based upon 5 times the expected half-life of dexamethasone) except patients who are taking steroids for physiological replacement or in the case of Inhaled or topical steroids or other immunosuppressive medications. If alternative corticosteroid therapy has been used, consultation with the PI is required to determine the washout period prior to initiating study treatment.

11. Major surgical procedure, open biopsy (excluding skin cancer resection), or significant traumatic injury within 14 days of initiating study drug (unless the wound has healed) or anticipation of the need for major surgery during the study.

12. Non-healing wound, ulcer, or bone fracture. 13. Women who are breast-feeding or pregnant. 14. Uncontrolled intercurrent illness (i.e., active infection ≥ grade 2) or concurrent condition that, in the opinion of the Investigator, would interfere with the study endpoints or the subject's ability to participate.

15. History of clinically significant cardiac disease or congestive heart failure > New York Heart Association (NYHA) class 2. Subjects must not have unstable angina (anginal symptoms at rest) or new-onset angina within the last 3 months or myocardial infarction within the past 6 months or a history of myocarditis. Also, • prior myocarditis of any etiology. • Left ventricular ejection fraction (LVEF) assessment with documented LVEF < 50% by either transthoracic echocardiogram (TTE) or multigated acquisition scan (TTE preferred test) within 6 months prior to the start of study treatment.

16. Troponin T (TnT) or I (TnI) > 2 × institutional ULN. Participants with TnT or TnI levels between > 1 to 2 × ULN will be permitted if repeat levels within 24 hours are ≤ 1 ULN. If TnT or TnI levels are between >1 to 2 × ULN within 24 hours, the participant may undergo a cardiac consultation and be considered for treatment, following cardiologist recommendation. When repeat levels within 24 hours are not available, a repeat test should be conducted as soon as possible. If TnT or TnI repeat levels beyond 24 hours are < 2 × ULN, the participant may undergo a cardiac consultation and be considered for treatment, following cardiologist recommendation. Notification of the decision to enroll the participant following cardiologist recommendation has to be made to the principal investigator.

17. Investigational drug use within 14 days (or 5 half-lives, whichever is shorter) of the first dose of the triplet therapy.

18. The use of herbal supplements within 7 days. 19. History of non-infectious pneumonitis that required steroids or current pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2030-08-16 (Estimated); Study Completion 2032-08-16 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Hussein Tawbi, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org